CLINICAL TRIAL: NCT04485039
Title: A Post-Marketing Open-Label, 5 Period Crossover, Drug-Drug Interaction Study of Orally Adminstered TPOXX When Co-administered With 4 Different Phosphate Binders in Healthy Subjects
Brief Title: Drug-drug Interaction Study of TPOXX When Co-administered With Phosphate Binders
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: SIGA Technologies (Industry)
Collaborators: Biomedical Advanced Research and Development Authority (U.S. Federal Agency); PPD Development, LP (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Other
Other Study IDs: SIGA-246-023
Record Dates: First submitted 2020-05-11; First posted 2020-07-24 (Actual); Results first posted 2024-10-09 (Actual); Last update posted 2024-12-27 (Actual); Status verified 2024-12

CONDITIONS: Smallpox
MeSH Terms: conditions — Smallpox | interventions — tecovirimat; Sevelamer; sucroferric oxyhydroxide; calcium acetate; lanthanum carbonate

STUDY DESIGN:
Intervention Model Description: 5 period crossover
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (5):
- TPOXX: oral antiviral (Other): Single oral dose of TPOXX 600 mg
  Interventions: Drug: Tecovirimat
- TPOXX: oral antiviral and sevelamer carbonate (Other): Single oral dose of TPOXX 600 mg co-administered with single oral dose of 1600 mg sevelamer carbonate
  Interventions: Drug: Tecovirimat; Drug: sevelamer carbonate oral tablet
- TPOXX: oral antiviral and sucroferric oxyhydroxide (Other): Single oral dose of TPOXX 600 mg co-administered with single oral dose of 500 mg sucroferric oxyhydroxide chewable tablet
  Interventions: Drug: Tecovirimat; Drug: sucroferric oxyhydroxide chewable tablet
- TPOXX: oral antiviral and calcium acetate (Other): Single oral dose of TPOXX 600 mg co-administered with a single oral dose of 1334 mg calcium acetate
  Interventions: Drug: Tecovirimat; Drug: calcium acetate oral tablet
- TPOXX: oral antiviral and lanthanum carbonate (Other): Single oral dose of TPOXX 600 mg co-administered with a single oral dose of 500 mg lanthanum carbonate chewable tablet
  Interventions: Drug: Tecovirimat; Drug: Lanthanum Carbonate Chewable Tablet

INTERVENTIONS:
Drug: Tecovirimat — oral antiviral
  Other Names: TPOXX
Drug: sevelamer carbonate oral tablet — phosphate binder
  Other Names: Renvela
  Arms: TPOXX: oral antiviral and sevelamer carbonate
Drug: sucroferric oxyhydroxide chewable tablet — phosphate binder
  Other Names: Velphoro
  Arms: TPOXX: oral antiviral and sucroferric oxyhydroxide
Drug: calcium acetate oral tablet — phosphate binder
  Other Names: PhosLo
  Arms: TPOXX: oral antiviral and calcium acetate
Drug: Lanthanum Carbonate Chewable Tablet — phosphate binder
  Other Names: Fosrenol
  Arms: TPOXX: oral antiviral and lanthanum carbonate

SUMMARY:
An open-label, drug-drug interaction study with TPOXX and phosphate binders.

DETAILED DESCRIPTION:
A postmarketing open-label, 5 period crossover, drug-drug interaction study of orally administered TPOXX when coadministered with 4 different phosphate binders in healthy adult subjects.

ELIGIBILITY:
Inclusion Criteria:

* Each subject must meet all of the following criteria to be enrolled in this study:

  1. Subject is male or female 18 to 50 years of age, inclusive.
  2. Phosphorus levels within normal laboratory reference range.
  3. Women of childbearing potential have a negative human chorionic gonadotropin pregnancy test (serum) at the screening visit and a confirmatory negative serum pregnancy test on Day -1 of each period before receipt of study drug, and meet one of the following criteria:

     1. The subject or their partner has undergone surgical sterilization
     2. The subject is postmenopausal, defined as 12 consecutive months with no menses without an alternative medical cause and has a documented plasma follicle-stimulating hormone level >40 IU/mL

Exclusion Criteria:

Subjects meeting any of the following criteria will be excluded from the study:

1. Subject is a female who is pregnant or breastfeeding or planning to become pregnant within 3 months after the last dose of study drug.
2. Subject has a history of any clinically significant conditions including:

   * Asthma treated with oral systemic steroids within the past 6 months
   * Diabetes mellitus (type 1 or 2), with the exception of gestational diabetes
   * Hypertension that is poorly controlled (repeat readings >140 mm Hg systolic and/or >90 mm Hg diastolic)
   * Thyroidectomy or thyroid disease that required medication within the past 12 months
   * Serious angioedema episodes within the previous 3 years or requiring medication in the previous 2 years
   * Head trauma resulting in a diagnosis of traumatic brain injury other than concussion
   * Frequent episodes of headache.
3. Subject has received treatment in another clinical study of an investigational drug (or medical device) within 30 days or 5 half-lives (whichever is longer) before the first dose of study drug.
4. Subject has a history of relevant drug and/or food allergies (ie, allergy to TPOXX or excipients, or any significant food allergy that could preclude a standard diet in the study site).
5. Subject has any condition possibly affecting drug absorption (eg, previous surgery on the gastrointestinal tract, including removal of parts of the stomach, bowel, liver, gallbladder, or pancreas, with the exception of appendectomy).
6. Subject has evidence or history of clinically significant allergic (except for untreated, asymptomatic, seasonal allergies at time of the first dose of study drug), hematological, endocrine, pulmonary, gastrointestinal, cardiovascular, hepatic, psychiatric, or neurological disease. Exceptions to these criteria (eg, stable, mild joint disease unassociated with collagen vascular disease) may be made following discussions with the medical monitor.
7. Subject has a history of cardiac disease, symptomatic or asymptomatic arrhythmias, syncopal episodes, or risk factors for torsades de pointes (eg, heart failure, hypokalemia).
8. Subject has a family history of sudden cardiac death not clearly due to acute myocardial infarction.
9. Subject has a seizure disorder or history of seizures (does not include childhood febrile seizures) or a past history that increases seizure risks such as significant head injury that caused loss of consciousness or other changes in the subject's daily function, concussion, stroke, central nervous system infection or disease, or alcohol or drug abuse or family history of idiopathic seizures.
10. Subject has a history of a peptic ulcer or significant gastrointestinal bleeding.
11. Subject has a bleeding disorder diagnosed by a doctor (eg, factor deficiency, coagulopathy, or platelet disorder requiring special precautions) or significant bruising or bleeding difficulties with blood draws.
12. Subject has a malignancy that is active, or treated malignancy for which there is not reasonable assurance of sustained cure, or malignancy that is likely to recur during the period of the study (subject should be in complete remission for at least 5 years).
13. Subject has neutropenia or other blood dyscrasia determined to be clinically significant by the investigator.
14. Subject has used any of the following prohibited medications from within 7 days (or 5 half lives, whichever is longer) before the first dose of study drug: antidiabetic medication; anticoagulants; anticonvulsants; substrates of the breast cancer resistance protein transporter including methotrexate, mitoxantrone, imatinib, irinotecan, lapatinib, rosuvastatin, sulfasalazine, and topotecan; substrates of CYP2C8 including repaglinide, paclitaxel, Montelukast, pioglitazone, rosiglitazone; and substrates of CYP2C19 including S-mephenytoin, clobazam, diazepam, rabeprazole, voriconazole, lansoprazole, and omeprazole. Medications not listed here that are known (or thought) to be CYP3A4 substrates may be allowed at the investigator's discretion, after consultation with the medical monitor, if administration poses little to no risk to the subject.
15. Subject has a history of drug or alcohol abuse or dependency within the last year before screening.
16. Subject has a current or recent (<30 days before screening) history of clinically significant bacterial, fungal, or mycobacterial infection.
17. Subject has a current clinically significant viral infection.
18. Subject has a known clinically significant chronic viral infection (eg, human T cell lymphotropic virus I or II).
19. Subject has consumed grapefruit or grapefruit juice, Seville orange or Seville orange containing products (eg, marmalade), or caffeine- or xanthine containing products within 48 hours before the first dose of study drug.
20. Subject has used any prescription (excluding hormonal birth control) or over the counter medication (including herbal or nutritional supplements) within 14 days before the first dose of study drug.
21. Subject demonstrates long-term use (≥14 consecutive days) of glucocorticoids including oral or parenteral prednisone or equivalent (>20 mg total dose per day) or high-dose inhaled steroids (>800 mcg/day of beclomethasone dipropionate or equivalent) within the preceding 1 month (low-dose [≤800 mcg/day of beclomethasone dipropionate or equivalent] inhaled and topical steroids are allowed).
22. Subject has donated >450 mL blood or blood components within 30 days before the first dose of study drug. The investigator should instruct subjects who participate in this study to not donate blood or blood components for 4 weeks after the completion of the study.
23. Subject is a smoker or has used nicotine or nicotine containing products (eg, cigarettes, electronic vapor cigarettes, cigars, chewing tobacco, snuff, nicotine patches, or nicotine gum) within 6 months before the first dose of study drug.
24. Subject has consumed pomegranate or pomegranate juice, pomelo fruits or pomelo juice, or alcohol within 72 hours before the first dose of study drug.
25. Subject reports participation in strenuous activity or contact sports within 24 hours before the first dose of study drug.
26. Subject has known hepatitis B or C infection or positive test for hepatitis B surface antigen, hepatitis C virus antibody, or human immunodeficiency virus type 1 or 2 antibodies at screening.
27. Subject has a positive test result for amphetamines (including methamphetamines and ecstasy/methylenedioxymethamphetamine), barbiturates, benzodiazepines, cannabinoids (including tetrahydrocannabinol), cocaine metabolites, opiates (including heroin, codeine, and oxycodone), or alcohol at screening or check-in.
28. Subject has any of the following laboratory test results within 28 days before the first dose of study drug:

    * Estimated serum creatinine clearance (Cockcroft-Gault) <70 mL/min
    * Creatinine in males >1.7 mg/dL and in females >1.4 mg/dL (1.3 times the upper laboratory reference range)
    * Hemoglobin ≤10% of the lower laboratory reference range
    * White blood cell count considered to be clinically significant by the investigator
    * Absolute neutrophil count <1000 cells/mm3
    * Platelets not within ±10% of laboratory reference range
    * Alanine aminotransferase >2.0 times above the upper laboratory reference range
    * Aspartate aminotransferase >2.0 times above the upper laboratory reference range
    * Alkaline phosphatase >20% above the upper laboratory reference range
    * Hemoglobin A1c ≥7.0%
    * Cholesterol ≥300 mg/dL and low density lipoprotein ≥190 mg/dL.
29. Subject has a blood pressure considered to be clinically significant by the investigator. Blood pressure may be retested twice in the sitting position at 5 minute intervals.
30. Subject has a resting heart rate of <40 beats per minute or >110 beats per minute at screening.
31. Subject has an abnormal ECG at screening that is determined by the investigator to be clinically significant.
32. Male subject has a QT interval corrected using Fridericia's formula (QTcF) >450 ms or female subject has a QTcF >470 ms at screening or Day -1.
33. In the opinion of the investigator, the subject is not suitable for entry into the study.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 44 (Actual)
Dates: Start 2022-06-08 (Actual); Primary Completion 2022-12-15 (Actual); Study Completion 2023-04-23 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Dennis Hruby, PhD, Study Director — SIGA Technologies Chief Scientific Officer
Locations (1):
- PPD Phase I Clinic, Austin, Texas, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- TPOXX Co-administered With Phosphate Binders: Single oral dose of TPOXX 600 mg, followed by TPOXX co-administered with a single oral dose of each of the following four phosphate binders individually with washout between each period:
  sevelamer carbonate 1600 mg sucroferric oxyhydroxide chewable tablet 500 mg calcium acetate 1334 mg lanthanum carbonate chewable tablet 500 mg
  Participants were randomly assigned to receive TPOXX with one of each of the phosphate binders in 1:1:1:1 ratio to maintain enrollment across all periods. The order of administration of TPOXX with each individual phosphate binder had no bearing on study design due to washout between periods.
Period: TPOXX Only
Arm/Group | TPOXX Co-administered With Phosphate Binders
Started | 44
Completed | 41
Not Completed | 3
Not completed — Adverse Event | 2
Not completed — Physician Decision | 1
Period: TPOXX With Sevelamer Carbonate
Arm/Group | TPOXX Co-administered With Phosphate Binders
Started | 41
Completed | 39
Not Completed | 2
Not completed — Adverse Event | 1
Not completed — Withdrawal by Subject | 1
Period: TPOXX With Sucroferric Oxyhydroxide
Arm/Group | TPOXX Co-administered With Phosphate Binders
Started | 39
Completed | 39
Not Completed | 0
Period: TPOXX With Calcium Acetate
Arm/Group | TPOXX Co-administered With Phosphate Binders
Started | 39
Completed | 39
Not Completed | 0
Period: TPOXX With Lanthanum Carbonate
Arm/Group | TPOXX Co-administered With Phosphate Binders
Started | 39
Completed | 39
Not Completed | 0

BASELINE CHARACTERISTICS:
Groups:
- TPOXX: Oral Antiviral and Phosphate Binders: Single oral dose of TPOXX 600 mg co-administered with single oral dose of 1600 mg sevelamer carbonate Single oral dose of TPOXX 600 mg co-administered with single oral dose of 500 mg sucroferric oxyhydroxide chewable tablet Single oral dose of TPOXX 600 mg co-administered with a single oral dose of 1334 mg calcium acetate Single oral dose of TPOXX 600 mg co-administered with a single oral dose of 500 mg lanthanum carbonate chewable tablet.
Arm/Group | TPOXX: Oral Antiviral and Phosphate Binders
Number analyzed (Participants) | 44
Age, Customized [Mean (Standard Deviation); unit: years]
  Age | 33.5 (8.61)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 17
  Male | 27
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 16
  Not Hispanic or Latino | 28
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 21
  White | 22
  More than one race | 1
  Unknown or Not Reported | 0
Height (cm) [Mean (Standard Deviation); unit: centimeters] | 170.39 (8.674)
Weight (kg) [Mean (Standard Deviation); unit: kilograms] | 84.51 (18.012)
Body Mass Index (kg/m2) [Mean (Standard Deviation); unit: Kilograms Per Square Meter] | 29.10 (5.898)

OUTCOME MEASURES:

1. Primary Outcome: AUC0-inf
Description: Area under the plasma concentration of vs. time curve (AUC) of TPOXX from 0 extrapolated to infinity
Time Frame: Day 3
Population: healthy participants
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng*h/mL
Groups:
- TPOXX: Oral Antiviral Coadministered With Sevelamer Carbonate: A single oral dose of 600 mg TPOXX coadministered with a single oral dose of 1600 mg sevelamer carbonate
- TPOXX: Oral Antiviral Coadministered With Sucroferric Oxyhydroxide: A single oral dose of 600 mg TPOXX coadministered with a single oral dose of 500 mg sucroferric oxyhydroxide chewable tablet
- TPOXX: Oral Antiviral Coadministered With Calcium Acetate: A single oral dose of 600 mg TPOXX coadministered with a single oral dose of 1334 mg calcium acetate
- TPOXX: Oral Antiviral Coadministered With Lanthanum Carbonate: A single oral dose of 600 mg TPOXX coadministered with a single oral dose of 500 mg lanthanum carbonate chewable tablet
Arm/Group | TPOXX: Oral Antiviral | TPOXX: Oral Antiviral Coadministered With Sevelamer Carbonate | TPOXX: Oral Antiviral Coadministered With Sucroferric Oxyhydroxide | TPOXX: Oral Antiviral Coadministered With Calcium Acetate | TPOXX: Oral Antiviral Coadministered With Lanthanum Carbonate
Number analyzed (Participants) | 44 | 41 | 39 | 39 | 39
ng*h/mL | 16300 (39.6) | 21600 (46.4) | 21000 (37.8) | 19500 (37.4) | 21000 (25.9)

2. Primary Outcome: Cmax
Description: Cmax - maximum observed plasma concentration of TPOXX
Time Frame: Day 3
Population: healthy participants
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | TPOXX: Oral Antiviral | TPOXX: Oral Antiviral Coadministered With Sevelamer Carbonate | TPOXX: Oral Antiviral Coadministered With Sucroferric Oxyhydroxide | TPOXX: Oral Antiviral Coadministered With Calcium Acetate | TPOXX: Oral Antiviral Coadministered With Lanthanum Carbonate
Number analyzed (Participants) | 44 | 41 | 39 | 39 | 39
ng/mL | 1230 (29.5) | 1440 (29.6) | 1440 (32.7) | 1370 (32.0) | 1510 (26.1)

3. Secondary Outcome: Adverse Events
Description: Number of participants with adverse events when TPOXX is coadministered with phosphate binders
Time Frame: 59 days
Population: Healthy participants
Measure: Number; unit: participants
Groups:
- TPOXX: Oral Antiviral Coadministered With: A single oral dose of 600 mg TPOXX coadministered with a single oral dose of 500 mg sucroferric oxyhydroxide chewable tablet.
- TPOXX: Oral Antiviral Coadministered With Lanthanum Carbonate: single oral dose of 600 mg TPOXX coadministered with a single oral dose of 500 mg lanthanum carbonate chewable tablet
Arm/Group | TPOXX: Oral Antiviral | TPOXX: Oral Antiviral Coadministered With Sevelamer Carbonate | TPOXX: Oral Antiviral Coadministered With | TPOXX: Oral Antiviral Coadministered With Calcium Acetate | TPOXX: Oral Antiviral Coadministered With Lanthanum Carbonate
Number analyzed (Participants) | 44 | 41 | 39 | 39 | 39
participants | 6 | 7 | 7 | 3 | 2

ADVERSE EVENTS:
Time Frame: Adverse event data was collected from Day 1 though the Day 59 follow-up telephone call. All AEs were followed until stable or until resolution as determined by the investigator and/or medical monitor.
Description: All-Cause Mortality was not assessed
Arm/Group | TPOXX: Oral Antiviral | TPOXX: Oral Antiviral and Sevelamer Carbonate | TPOXX: Oral Antiviral and Sucroferric Oxyhydroxide | TPOXX: Oral Antiviral and Calcium Acetate | TPOXX: Oral Antiviral and Lanthanum Carbonate
All-Cause Mortality (participants affected / at risk) | 0/0 | 0/0 | 0/0 | 0/0 | 0/0
Serious Adverse Events (participants affected / at risk) | 1/44 | 0/41 | 0/39 | 0/39 | 0/39
Other Adverse Events (participants affected / at risk) | 6/44 | 7/41 | 7/39 | 3/39 | 2/39
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | TPOXX: Oral Antiviral (N=44) | TPOXX: Oral Antiviral and Sevelamer Carbonate (N=41) | TPOXX: Oral Antiviral and Sucroferric Oxyhydroxide (N=39) | TPOXX: Oral Antiviral and Calcium Acetate (N=39) | TPOXX: Oral Antiviral and Lanthanum Carbonate (N=39)
Urinary tract infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | TPOXX: Oral Antiviral (N=44) | TPOXX: Oral Antiviral and Sevelamer Carbonate (N=41) | TPOXX: Oral Antiviral and Sucroferric Oxyhydroxide (N=39) | TPOXX: Oral Antiviral and Calcium Acetate (N=39) | TPOXX: Oral Antiviral and Lanthanum Carbonate (N=39)
Headache (Nervous system disorders) | 2 (2) | 2 (2) | 2 (2) | 3 (3) | 1 (1)
Dizziness (Nervous system disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Somnolence (Nervous system disorders) | 1 (1) | 1 (1) | 1 (1) | 1 (1) | 0 (0)
Nausea (Gastrointestinal disorders) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 1 (1)
Vomiting (Gastrointestinal disorders) | 1 (1) | 1 (1) | 1 (1) | 1 (1) | 0 (0)
Abdominal Discomfort (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 1 (1)
Diarrhoea (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dry mouth (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Myalgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Fatigue (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Feeling hot (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Tinea pedis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Bum oral cavity (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Concussion (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Acne (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pruritus (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Skin irritation (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Eyelid irritation (Eye disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
SARS-CoV-2 test positive (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Nervousness (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Dysmenorrhoea (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Physical assault (Social circumstances) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The agreement restricts the right of the PI to discuss or publish trial results.

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2023-06-28): https://cdn.clinicaltrials.gov/large-docs/39/NCT04485039/Prot_SAP_001.pdf